CLINICAL TRIAL: NCT03067298
Title: Prediction of Preeclampsia and Other Pregnancy Complications Following Combined Iterative Screening
Acronym: PREDICTION2
Status: Completed | Type: Observational
Sponsor: Emmanuel Bujold (Other)
Collaborators: Thermo Fisher Scientific, Inc (Industry); Laval University (Other)
Responsible Party: Sponsor-Investigator, Emmanuel Bujold, MD, FRCSC, CHU de Quebec-Universite Laval
Organization: CHU de Quebec-Universite Laval (Other)
Other Study IDs: 2017-3219
Record Dates: First submitted 2017-01-18; First posted 2017-03-01 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Preeclampsia; Preterm Birth; Fetal Growth Restriction; Intra Uterine Fetal Death
Keywords: pregnancy; screening; doppler; markers; PlGF; sFlt-1; placenta
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — maternal serum, maternal plasma (cell-free DNA), maternal urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Preterm birth (PTB), preeclampsia (PE), fetal growth restriction (FGR) and intra-uterine fetal death (IUFD) constitutes the main causes of perinatal morbidity and mortality and are called "Great Obstetrical Syndromes". Algorithms to predict those outcomes have been developed by combining maternal characteristics (history, age, BMI, blood pressure), biochemical (sFlt-1, β-hCG, PlGF, AFP) and sonographic (uterine artery Doppler, 3D of placenta, cervical length, nasal bone measurement, nuchal translucency) markers. Another prospective observational study ("PREDICTION study" NCT 02189148) is also ongoing, which aims to validate those algorithms at the first trimester of pregnancy.

Recent data suggest that repeating the same measurements later in pregnancy could improve the detection rates, allowing closer monitoring of high-risk patients and potential therapeutics under investigation. The current study (PREDICTION2) is an ancillary study of PREDICTION and aims at validating the use of these markers in a combined iterative manner in the prediction of preeclampsia and other obstetrical outcomes.

DETAILED DESCRIPTION:
The objective of this study is to validate the predictive values of biophysical (maternal blood pressure); biochemical (sFlt-1, β-hCG, PlGF, and AFP) and ultrasonographic (cervical length, Doppler, 3D evaluation of the placenta, 3D nasal bone) biomarkers at several timepoints for the prediction of adverse pregnancy outcomes including preterm birth, preeclampsia, fetal growth restriction and intra-uterine fetal death.

These biomarkers will be evaluated at 14-16 weeks, 20-24 weeks and 30-34 weeks. Those specific gestational ages have been selected because they correspond to the typical clinical/hospital visits for prenatal blood and/or ultrasound screening.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous pregnant women participating in Prediction study (NCT02189148)

Exclusion Criteria:

* <18 years old at recruitment;
* multiple pregnancies;
* fetal congenital malformation;
* positive for HIV or hepatitis C;
* fetal demise at recruitment;
* women planning a delivery outside the participating hospitals;
* women not able to provide an informed consent to the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 805 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
preeclampsia | >20 weeks of preeclampsia
  1) de novo hypertension with systolic blood pressure ≥ 140 mmHg or diastolic blood pressure >90 mmHg on two occasions at least four hours apart, after 20 weeks of pregnancy, and 2) associated with proteinuria ≥300 mg/24 h or at least '2 +' protein on urine dipstick or an adverse conditions

SECONDARY OUTCOMES:
Fetal growth restriction | neonatal weight at birth (on the day of birth)
  defined as a birth weight below the 10th centile (or below the 3rd centile for severe FGR) of Canadian reference growth charts.
Preterm birth | between 20-37 weeks of gestation
  defined as delivery <37 weeks of gestation.
Intra uterine fetal death | from the 20th week of gestation to the moment of birth
  fetal death during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bujold, MD, MSc, Principal Investigator — CHU de Quebec
Locations (1):
- CHU de Quebec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No